CLINICAL TRIAL: NCT04185870
Title: Optical Surface Imaging Versus Conventional Photography as a Tool to Document the Surface Geometry of Pectus Excavatum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: METCZ20190151
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Pectus Excavatum; Funnel Chest
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Intervention Model Description: All participants will receive standard photographs and a 3D scan
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D scan and standard photography arm (Experimental): All participants will receive a 360 degrees 3D scan of their chest/pectus excavatum. In addition, all participants will receive a the standard photographs and specialised recordings of the current work-up to document their chest/pectus excavatum.
  Interventions: Diagnostic Test: 3D scan; Diagnostic Test: Standard photography

INTERVENTIONS:
Diagnostic Test: 3D scan — All participants will receive a 360 degrees 3D scan of their chest/pectus excavatum.
Diagnostic Test: Standard photography — All participants will receive a the standard photographs and specialised recordings of the current work-up to document their chest/pectus excavatum.

SUMMARY:
Pectus excavatum is the most common congenital anterior chest wall deformity, known to occur in 1:400 of new-borns. Complaints may be of cosmetic nature or as a consequence of (cardio)pulmonary impairment. Part of the current work-up of pectus excavatum patients in Zuyderland Medical Centre (Heerlen, the Netherlands) is visual documentation of the deformity. Visual documentation is performed utilising a single-reflex camera and consists of 5 standard photographs (acquired from different angles) and two specialised recordings. These specialised recordings encompass a recording to measure the pectus excavatum's depth and a raster stereography recording to create a three-dimensional perspective. However, this form of visual documentation is not efficient, as it is time- and labor-intensive for the photographer and patient.

Recently, another study started that aims to investigate whether three-dimensional (3D) optical surface scans can be used to determine pectus severity, as compared to chest radiographs and computed tomography scans (3DPECTUS study; METCZ20190048; NCT03926078). Building on this study it was determined whether 3D optical surface scans can be used as a tool to document the surface geometry of pectus excavatum. To determine whether the current standard photographs and specialised recordings can be replaced by a 3D scan, both methods are compared. To make this comparison, the pectus excavatum depth was chosen as an objective measure of agreement. If there is good agreement, it is assumed that the standard photos can be replaced by a 3D photo in the current work-up. This will subsequently result in a time saving as well as a reduced burden for the patient while acquisition of 3D scans takes only 10 seconds.

ELIGIBILITY:
Inclusion Criteria:

* All participants of the 3D PECTUS study (METCZ20190048; NCT03926078) that received a 3D scan and standard photographies.

Exclusion Criteria:

* Participants in which the photography based pectus excavatum depth was measured in the transversal plane.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Standard photography based pectus excavatum depth | 2 months
  The pectus excavatum depth is derived from one of the specialized recordings. The depth is obtained by placing a rigid bar with rule over the most excavated part in the transversal plane.
3D scan based pectus excavatum depth | 2 months
  The pectus excavatum depth is calculated by slicing the 3D scan in the longitudinal direction. The pectus depth is subsequently calculated from the transversal slice with the most severe excavation.
Absolute agreement between the 3D scan and photography based pectus excavatum depth. | 2 months
  The absolute agreement was assessed by calculation of the intraclass correlation coefficient.

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medical Centre, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Daemen JHT, Loonen TGJ, Coorens NA, Maessen JG, Maal TJJ, Hulsewe KWE, Vissers YLJ, de Loos ER. Photographic documentation and severity quantification of pectus excavatum through three-dimensional optical surface imaging. J Vis Commun Med. 2020 Oct;43(4):190-197. doi: 10.1080/17453054.2020.1784711. Epub 2020 Aug 14. PMID 32791868